CLINICAL TRIAL: NCT01520324
Title: Intraepithelial Neoplasia Detection Rate After Single Oral Dose of Methylene Blue MMX Modified Release Tablets Administered to Patients With Long Standing Ulcerative Colitis Undergoing Colonoscopy.
Brief Title: Neoplasia Detection With Methylene Blue MMX Tablets in Patients With UC Undergoing Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CB-17-01/04
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with UC undergoing colonoscopy (Experimental)
  Interventions: Device: oral delivery mucosal stain

INTERVENTIONS:
Device: oral delivery mucosal stain — 200mg methylene blue MMX tablet taken prior to colonoscopy

SUMMARY:
Evaluation of the intraepithelial neoplasia detection rate in patients with long standing ulcerative colitis undergoing mucosal staining with oral methylene blue MMX tablets prior to colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* endoscopically verified UC signed written informed consent

Exclusion Criteria:

* Known or suspected GI obstruction or perforation Liver or renal impairment, malignancy, pregnancy or lactation, suppressed PT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, MD, Principal Investigator — Humanitas Hospital, Italy
Locations (1):
- Centre for Research & Care of Intestinal Diseases, Rozzano, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients with a diagnosis of ulcerative colitis dating not less than 8 years.
Pre-assignment Details: This was an exploratory, non-comparative study with no randomization. All subjects were allocated to receive Selg 1000® 4 L bowel preparation, the day before colonoscopy. All study subjects were allocated to receive 200 mg of Methylene Blue MMX® tablets during and at the end of the intake of bowel cleansing preparation.
Period: Overall Study
Arm/Group | Patients With UC Undergoing Colonoscopy
Started | 53
Completed | 52
Not Completed | 1
Not completed — Subject discontinued (moderate illness) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With UC Undergoing Colonoscopy
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] — 18 <= age years
  Years
    Age | 45.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 168.9 (8.4)
Body weight [Mean (Standard Deviation); unit: kg] | 70.04 (9.57)

OUTCOME MEASURES:

1. Primary Outcome: Detected Intraepithelial Neoplasia
Description: Rate of intraepithelial neoplasiae detection in the whole colon.
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Mean (Standard Deviation); unit: Number of detected IN
Groups:
- Full Analysis Set (FAS): All enrolled subjects, who received at least one dose of the test investigational medicinal product and had at least one evaluation of the number of detected neoplasiae.
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
Number of detected IN | 0.2 (0.5)
Statistical Analysis 1: Comparison: Full Analysis Set (FAS); The number of detected neoplasiae for each patient was listed and summarised by descriptive statistics. Number and percentage of patients with intraepithelial neoplasiae was presented; Test type: Other — The data documented in this trial and the parameters measured were described using classic statistics, i.e. mean, SD, CV(%), median, minimum and maximum values for quantitative variables and frequencies for qualitative variables; The data documented in this trial and the parameters measured were described using classic statistics, i.e. mean, SD, CV(%), median, minimum and maximum values for quantitative variables and frequencies for qualitative variables

2. Primary Outcome: Intraepithelial Neoplasia (IN) Detection Rate (True Positive Findings)
Description: The rate of intraepithelial neoplasiae detection in the whole colon is summarised along with the number and percentage of subjects affected. The number and percentage of false and true negative and of false and true positive findings of intraepithelial neoplasiae are also listed.
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Number; unit: percentage of true pos. findings of IN
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
percentage of true pos. findings of IN | 7.7

3. Primary Outcome: Intraepithelial Neoplasia (IN) Detection Rate (False Positive Findings)
Description: as for outcome 2
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Number; unit: percentage of false pos. findings of IN
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
percentage of false pos. findings of IN | 7.7

4. Primary Outcome: Intraepithelial Neoplasia (IN) Detection Rate (True Negative Findings)
Description: as for outcome 2
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Number; unit: percentage of true neg. findings of IN
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
percentage of true neg. findings of IN | 78.8

5. Primary Outcome: Intraepithelial Neoplasia (IN) Detection Rate (False Negative Findings)
Description: as for outcome 2
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Number; unit: percentage of false neg. findings of IN
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
percentage of false neg. findings of IN | 5.8

6. Secondary Outcome: The Extent and Severity of the Inflamed Mucosa
Description: The inflammation conditions of the mucosa were evaluated during the colonoscopy and, afterwards, in the bioptic specimens.
  Rachmilewitz EI and Saverymuttu scores were used to assess inflammation. Rachmilewitz's scoring system for endoscopic index (EI) measures granulation scattering reflected light, vascular pattern, vulnerability of mucose and mucosal damage on a scoring scale of 0 to 4 from normal to damaged.
  Saverymuttu's scoring system for enteric specimens assesses disease activity in the bowel by rating histological changes in enterocytes, crypts, lamina propria mononuclear cells and lamina propria neutrophils.
  The average score for histological changes in individual biopsy specimens was summed and converted into a grade from 1 to 4, increasing in severity.
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Mean (Standard Deviation); unit: Rachmilewitz and Saverymuttu scores
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
Rachmilewitz and Saverymuttu scores
  Rachmilewitz EI | 2.1 (3.0)
  Saverymuttu grade | 1.1 (1.0)

7. Secondary Outcome: The Mucosal Staining Efficacy of Methylene Blue MMX® Tablets After a Total Oral Dose of 200 mg Administered During and at the End of the Intake of the Bowel Cleansing Preparation.
Description: The mucosal staining efficacy of Methylene Blue MMX® tablets was assessed in all 4 examined colonic regions (ascending, transverse and descending colon and rectosigmoid).
  The staining efficacy in each colon region was assessed scoring the observed staining percentage as reported below:
  0. no staining
  1. traces (poor traces in colon mucosa)
  2. detectable (at least the 25% of colon mucosa is stained)
  3. acceptable (at least the 50% of colon mucosa is stained)
  4. good (at least the 75% of colon mucosa is stained)
  5. overstained (the 100% of the colon mucosa is over stained)
Time Frame: During colonscopy (usually <15 min) and subsequent histological analysis
Measure: Mean (Standard Deviation); unit: Staining score
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
Staining score
  Ascending colon | 3.4 (1.0)
  Transverse colon | 3.0 (0.9)
  Descending colon | 2.9 (1.1)
  Rectosigmoid | 2.8 (1.1)

8. Secondary Outcome: Bowel Cleansing Quality Evaluated by Boston Bowel Preparation Scale After Intake of Bowel Cleansing Formulation and of a Total Dose of 200 mg of Methylene Blue MMX Tablets Administered During and at the End of the Intake of the Bowel Cleansing Formulation
Description: The Boston Bowel Preparation Score (BBPS) was used to rate colon cleansing quality. Each of the following 3 regions was rated: right, mid and rectosigmoid colon. The following 4-point scale (0-3) was used.
  0 - unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared
  1. - portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid
  2. - minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well
  3. - entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
  Each region of the colon received a "segment score" from 0 to 3 and these segment scores were summed for a total BBPS score ranging from 0 to 9. Therefore, the maximum BBPS score for a perfectly clean colon, without any residual liquid, is 9 and the minimum BBPS score for an unprepared colon is 0.
Time Frame: During colonscopy (usually <15 min)
Measure: Mean (Standard Deviation); unit: Boston bowel preparation scale (BBPS)
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 52
Boston bowel preparation scale (BBPS)
  Right colon | 1.3 (0.5)
  Mid colon | 1.7 (0.5)
  Rectosigmoid colon | 1.7 (0.5)

ADVERSE EVENTS:
Time Frame: On the day before colonoscopy (day 1), the subjects took the investigational product at home during the intake of the bowel cleansing preparation according to the given instructions. On the following day (day 2), the patients returned to the clinic for colonoscopy. The investigator inquired the subjects about occurrence of any AE and the intake of concomitant medications. It was over these two days the AEs were monitored.
Arm/Group | Full Analysis Set (FAS)
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 8/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Set (FAS) (N=53)
Nausea (Gastrointestinal disorders) | 8 (8) — Mild nausea for 6 subject s Moderate for 2 subjects
Vomiting (Gastrointestinal disorders) | 1 (1) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication to be reviewed by sponsor prior to submission.